CLINICAL TRIAL: NCT01754662
Title: A Pilot Study Investigating the Effects of the Combined Effects of Cocoa and Soy Polyphenols in a Soy Protein Matrix on Insulin Resistance and Cardiovascular Disease Risk in Type 2 Diabetes - A Randomised Placebo-Controlled Double-Blind Parallel Study
Brief Title: Effects of Combining Cocoa and Soy in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R1188
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes; Dietary Intervention
Keywords: Type 2 diabetes; Cardiovascular risk; Endothelial function; Insulin resistance; Soy; Isoflavones; Cocoa; Diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Soybean Proteins; Isoflavones; Chocolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Soy protein with isoflavones and cocoa (Experimental): Soy protein with isoflavones and cocoa bars. 2 bars daily for 8 weeks.
  Interventions: Dietary Supplement: Soy protein; Dietary Supplement: Isoflavones; Dietary Supplement: Cocoa
- Soy protein alone with cocoa (Experimental): Soy protein alone with cocoa with no isoflavones. 2 bars daily for 8 weeks.
  Interventions: Dietary Supplement: Soy protein; Dietary Supplement: Cocoa
- Soy protein with soy isoflavones (Experimental): Soy protein with isoflavones bar. 2 bars daily for 8 weeks.
  Interventions: Dietary Supplement: Soy protein; Dietary Supplement: Isoflavones
- Soy protein alone (Experimental): Soy protein alone without soy isoflavone or cocoa polyphenol. 2 bars daily for 8 weeks.
  Interventions: Dietary Supplement: Soy protein
- Placebo (Placebo Comparator): Placebo bar without soy protein, isoflavones or cocoa polyphenols. 2 bars daily for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soy protein — 2 bars daily for 8 weeks.
  Arms: Soy protein alone; Soy protein alone with cocoa; Soy protein with isoflavones and cocoa; Soy protein with soy isoflavones
Dietary Supplement: Isoflavones — 2 bars daily for 8 weeks.
  Arms: Soy protein with isoflavones and cocoa; Soy protein with soy isoflavones
Dietary Supplement: Cocoa — 2 bars daily for 8 weeks.
  Arms: Soy protein alone with cocoa; Soy protein with isoflavones and cocoa
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Diabetes is an increasingly common condition affecting millions of people world wide. The cornerstone of treatment is lifestyle that includes looking at the way how people eat. It is known that food containing compounds called polyphenols can reduce the risk of heart disease risk in people with diabetes. Two foods that are rich sources of polyphenols are cocoa (epicatechins) and soy (isoflavones). Previous studies have shown the benefits of these foods in the diets of people with diabetes. It has also been shown that soy isoflavones and cocoa polyphenols can improve the mood in certain groups of patients.

What is not known is whether there is any extra benefit of combining soy protein and isoflavones with cocoa.

The aim of the study is to look at the modification of cardiovascular risk by soy and/or cocoa in patients with type 2 diabetes, alone or in combination.

DETAILED DESCRIPTION:
1. General information about the study

   The target number of participants is 100. All participants are patients with type 2 diabetes on diet alone or metformin treatment. Participants will be asked to eat two soy bars daily for 8 weeks. The length of the study is 10 weeks and involves 4 visits at the Diabetes Research Centre in Hull, UK.

   The bars will contain:
   * soy protein alone, or
   * soy protein with additional isoflavones, or
   * soy protein with cocoa, or
   * soy protein with isoflavones and cocoa, or
   * placebo bars without soy protein, isoflavones or cocoa.

   The study is randomised (a computer based allocation schema will be used to decide which bars the participant will need to consume). Participants have the same 20% chance to be participant of any of the above groups. The study is placebo-controlled (there is one arm of placebo bars without soy protein, additional isoflavones or cocoa). The study is double-blind (neither the participants or the research team will know which bars they will take).
2. Study-specific procedures

Visit 1 (week 0). Non-fasting visit. Interested participants discuss the study with a member of the study team who will explain each aspect of the study, following which informed consent will be then obtained. Subsequently, blood pressure, weight, height and waist circumference will be measured, medical history and list of medication are recorded, and blood is taken to determine eligibility. A dietitian will explain about eating a normal diet and the foods we would like the participants to avoid during the study. Vegetarian patients may include too much soy in the diet and for this reason they will not be able to take part in the study. All participants will be non smokers.

Visit 2 (week 2)and Visit 4 (week 10). Fasting visits. Fasting blood is taken and the EndoPAT is performed. Weight, height and waist circumference measurement performed. The EndoPAT test takes between 20-30 minutes. The first box of study bars is dispensed during visit 2. Participants need to consume two bars daily. All remaining uneaten bars and empty wrappers will be collected during visit 4.

Visit 3 (week 6). Non-fasting visit. Height, weight, abdominal circumference, blood pressure are measured. Second box of study bars is dispensed.

Participants are asked to complete a one week food diary and a three day hunger questionnaire before the fasting blood tests. The food diary includes mood rating scales to assess the effect of the consumption of the bars on mood. Participants need to complete these prior to Visit 2 and visit 4.

Participants have 24 hours blood pressure measurement prior to Visit 2 and Visit 4.

24 hours urine collection also takes place prior to visit 2 and visit 4.

3. Optional test incorporated into the study: Body Volume Index measurement Based on participants preference, Body Volume Index measurement is offered as a complementary tool to assess body shape and weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes controlled by diet or metformin only
* Stable medication history for 3 months prior to screening visit
* Age 45-80

Exclusion Criteria:

* Patients with concurrent illness or any medication (especially antibiotics)3 months prior to enrollment that would effect the study results based on investigator's judgement
* Patients not wishing to allow disclosure to their GPs
* Pre-menopausal women or on hormone replacement therapy
* HbA1c >9% at screening
* Patients with known food allergies
* Smokers
* Vegans and vegetarians

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Insulin resistance, lipid profile | 8 weeks
  Soy with isoflavones and cocoa polyphenols have a greater impact on insulin resistance, lipid parameters in type 2 diabetes than seen with soy protein alone, soy protein with isoflavones and soy protein with cocoa polyphenols.

SECONDARY OUTCOMES:
Cardiovascular risk | 8 weeks
  Soy with isoflavones reduces cardiovascular risk as measured by fasting lipids and blood pressure
Isoflavones | 8 weeks
  Soy with isoflavones increases plasma isoflavones
Endothelial function | 8 weeks
  Soy and cocoa improves endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Atkin, Principal Investigator — University of Hull
Locations (1):
- Michael White Diabetes Centre, Hull, North Humberside, United Kingdom

REFERENCES:
- [Background] Anderson JW, Smith BM, Washnock CS. Cardiovascular and renal benefits of dry bean and soybean intake. Am J Clin Nutr. 1999 Sep;70(3 Suppl):464S-474S. doi: 10.1093/ajcn/70.3.464s. PMID 10479219
- [Background] Vedavanam K, Srijayanta S, O'Reilly J, Raman A, Wiseman H. Antioxidant action and potential antidiabetic properties of an isoflavonoid-containing soyabean phytochemical extract (SPE). Phytother Res. 1999 Nov;13(7):601-8. doi: 10.1002/(sici)1099-1573(199911)13:73.0.co;2-o. PMID 10548755
- [Background] Lee DS, Lee SH. Genistein, a soy isoflavone, is a potent alpha-glucosidase inhibitor. FEBS Lett. 2001 Jul 13;501(1):84-6. doi: 10.1016/s0014-5793(01)02631-x. PMID 11457461
- [Background] Sorenson RL, Brelje TC, Roth C. Effect of tyrosine kinase inhibitors on islets of Langerhans: evidence for tyrosine kinases in the regulation of insulin secretion. Endocrinology. 1994 Apr;134(4):1975-8. doi: 10.1210/endo.134.4.8137766.
- [Background] Wagner JD, Cefalu WT, Anthony MS, Litwak KN, Zhang L, Clarkson TB. Dietary soy protein and estrogen replacement therapy improve cardiovascular risk factors and decrease aortic cholesteryl ester content in ovariectomized cynomolgus monkeys. Metabolism. 1997 Jun;46(6):698-705. doi: 10.1016/s0026-0495(97)90016-0. PMID 9186308
- [Background] Duncan AM, Underhill KE, Xu X, Lavalleur J, Phipps WR, Kurzer MS. Modest hormonal effects of soy isoflavones in postmenopausal women. J Clin Endocrinol Metab. 1999 Oct;84(10):3479-84. doi: 10.1210/jcem.84.10.6067. PMID 10522983
- [Background] Goodman-Gruen D, Kritz-Silverstein D. Usual dietary isoflavone intake is associated with cardiovascular disease risk factors in postmenopausal women. J Nutr. 2001 Apr;131(4):1202-6. doi: 10.1093/jn/131.4.1202. PMID 11285326
- [Background] Hermansen K, Sondergaard M, Hoie L, Carstensen M, Brock B. Beneficial effects of a soy-based dietary supplement on lipid levels and cardiovascular risk markers in type 2 diabetic subjects. Diabetes Care. 2001 Feb;24(2):228-33. doi: 10.2337/diacare.24.2.228. PMID 11213870
- [Background] Tsai AC, Vinik AI, Lasichak A, Lo GS. Effects of soy polysaccharide on postprandial plasma glucose, insulin, glucagon, pancreatic polypeptide, somatostatin, and triglyceride in obese diabetic patients. Am J Clin Nutr. 1987 Mar;45(3):596-601. doi: 10.1093/ajcn/45.3.596. PMID 2881482
- [Background] Jayagopal V, Albertazzi P, Kilpatrick ES, Howarth EM, Jennings PE, Hepburn DA, Atkin SL. Beneficial effects of soy phytoestrogen intake in postmenopausal women with type 2 diabetes. Diabetes Care. 2002 Oct;25(10):1709-14. doi: 10.2337/diacare.25.10.1709. PMID 12351466
- [Background] Chedraui P, San Miguel G, Hidalgo L, Morocho N, Ross S. Effect of Trifolium pratense-derived isoflavones on the lipid profile of postmenopausal women with increased body mass index. Gynecol Endocrinol. 2008 Nov;24(11):620-4. doi: 10.1080/09513590802288283. PMID 19031218
- [Background] Scholey AB, French SJ, Morris PJ, Kennedy DO, Milne AL, Haskell CF. Consumption of cocoa flavanols results in acute improvements in mood and cognitive performance during sustained mental effort. J Psychopharmacol. 2010 Oct;24(10):1505-14. doi: 10.1177/0269881109106923. Epub 2009 Nov 26. PMID 19942640
- [Background] Konya J, Sathyapalan T, Kilpatrick ES, Atkin SL. The Effects of Soy Protein and Cocoa With or Without Isoflavones on Glycemic Control in Type 2 Diabetes. A Double-Blind, Randomized, Placebo-Controlled Study. Front Endocrinol (Lausanne). 2019 May 9;10:296. doi: 10.3389/fendo.2019.00296. eCollection 2019. PMID 31143160
- See also: publication link — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6521701/